CLINICAL TRIAL: NCT04774406
Title: Arterial Hypertension With PARP Inhibitors in Cancer Patients: an Observational and Retrospective Study Using the WHO Pharmacovigilance Database (ArteRIB)
Brief Title: Arterial Hypertension Related to PARP Inhibitors (ArteRIB)
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco 16022023
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — olaparib; rucaparib; niraparib; talazoparib; veliparib; pamiparib; fluzoparib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- parp inhibitors: All patients treated at least with 1 PARPi
  Interventions: Drug: olaparib, rucaparib, niraparib, talazoparib, veliparib, pamiparib, fluzoparib

INTERVENTIONS:
Drug: olaparib, rucaparib, niraparib, talazoparib, veliparib, pamiparib, fluzoparib — All patients treated at least with 1 PARPi (alone or in combination)

SUMMARY:
Although PARP inhibitors (PARPi) have proved effective in treating many cancers, few patients receiving PARPi may experience rare but serious (or not) adverse events such as hypertension whose data are scarce.

The objective was to investigate reports of hypertension related to PARPi, including olaparib, rucaparib, niraparib, talazoparib, veliparib, pamiparib, and fluzoparib using the World Health Organization's (WHO) pharmacovigilance database: VigiBase.

DETAILED DESCRIPTION:
Here, investigators use the World Health Organization's (WHO) database of individual safety case reports, to identify cases of hypertension AE related to PARPi.

ELIGIBILITY:
Inclusion Criteria:

* case reported in the World Health Organization (WHO) database (VigiBase) of individual safety case reports at the time of the extraction,
* patients treated with at least 1 PARPi (with ATC classification system): olaparib (ATC L01XX46), niraparib (ATC L01XX54), rucaparib (ATC L01XX55), talazoparib (ATC L01XX60), veliparib, pamiparib, fluzoparib (none).

Exclusion Criteria:

-chronology not compatible between the PARPi and adverse event

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients treated with PARPi and experiencing hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 2336 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
hypertension reports related to PARPi. | From inception to 16 Feb, 2023
  Identification of the hypertension adverse event related to PARP inhibitors reported in the World Health Organization's (WHO) database of individual safety case reports.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Joachim, Caen, Basse Normandie, France